CLINICAL TRIAL: NCT02364089
Title: Surgery of Subclinical Cortisol Secreting Adrenal Incidentalomas
Acronym: CHIRACIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2012/34
Record Dates: First submitted 2015-01-28; First posted 2015-02-16 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Adrenal Incidentalomas
Keywords: Adrenal Incidentaloma; Subclinical Cushing's syndrome; Hypertension; Cardiovascular Risk Factors; Metabolic Syndrome; Surgery of adrenal tumor
MeSH Terms: conditions — Adrenal incidentaloma; Hypertension; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery followed by intensive medical care (Experimental): Laparoscopic surgical removal of the adrenal tumor
  Interventions: Procedure: Laparoscopic surgical removal of the adrenal tumor
- Intensive medical treatment only (Active Comparator): Standardized medical treatment of hypertension by SAHR.
  Interventions: Drug: Standardized medical treatment of hypertension by SAHR

INTERVENTIONS:
Procedure: Laparoscopic surgical removal of the adrenal tumor
  Arms: Surgery followed by intensive medical care
Drug: Standardized medical treatment of hypertension by SAHR — Standardized anti-hypertensive drug regimen has been established according to international recommendations and includes the following steps:
  * step 1: Angiotensin converting enzyme inhibitor (ACE-I) or angiotensin II receptor antagonist (ARBs) at half-dose (Ranipril 5mg or Ibesartan 150 mg )
  * step 2: CEI or ARA2 at full dose (Ranipril 10 mg or Ibesartan 300 mg)
  * step 3: Add-on of Amlodipine 10 mg or Diltiazem LP 300 mg
  * step 4: Add-on of Indapamide LP 1.5 mg
  * step 5: Add-on of Spironolactone 25 mg
  * step 6: Add-on of Bisoprolol 10 mg
  * step 7: Add-on of Prazosine LP 5mg/day.
  Arms: Intensive medical treatment only

SUMMARY:
The general objective is to evaluate the consequences of surgical removal of SCSI on hypertension and cardiovascular risk factors in order to determine on an evidence-based basis if surgical excision of SCSI is preferable to an intensive medical regimen in patients with hypertension.

DETAILED DESCRIPTION:
Adrenal incidentalomas are unsuspected adrenal masses found during abdominal imaging. With the widespread use of computed tomography and MRI, adrenal incidentalomas are found in approximately 2% of patients. In an endocrinology setting, the majority of these masses are benign adenomas of the adrenal cortex. Approximately 10% of these adenomas display little excess of cortisol secretion associated to some degree of secretory autonomy but that are insufficient to generate overt Cushing's syndrome ("Subclinical Secreting Cortisol incidentalomas" or SCSI). However, hypertension and to a lesser degree obesity and impaired glucose tolerance are very frequent amongst patients with SCSI. The hypothesis that the mild hypercortisolism associated with SCSI is responsible for these clinical consequences is substantiated by few studies describing improvement after resection of SCSI. However, these studies were retrospective, uncontrolled and suffered from imprecision and numerous methodological bias. Thus, whether surgery is more beneficial than medical treatment is currently unknown and there is no consensus on the appropriate treatment for SCSI.

Patient selection Run-In period. Discontinuation of previous antihypertensive treatments and prescription of a standardized anti-hypertensive drug regimen (SAHR). Monthly Blood Pressure (BP) measurement using home BP monitoring. The duration of the Run-In periods will be ≤ 6 months and will end when BP will be controlled with the SAHR at two consecutive visits.

End of RI Second endocrine assessment for eligibility Randomization (Ra): 24h Ambulatory BP measurement, anthropometric and metabolic evaluation. Quality of life and cognition questionnaires. Randomization in 2 groups : Gr 1 Treatment group : Surgery followed by intensive medical care ; Gr 2 : Control Group : intensive medical care only.

Ra + 1Mo: Surgery in Group 1 Ra + 2.5 Mo to Ra + 13 Mo: 6 weeks interval follow-up Evaluation of home BP monitoring and adaptation of the SAHR. A step by step reduction of the SAHR will be attempted in the two patient groups at Ra+2.5Mo. A second attempt will systematically be performed in both groups at Ra+8.5 Medical evaluation of associated metabolic conditions (obesity, diabetes, dyslipidemia) and adaptation of treatments Record of medical events and side effects of treatments Ra + 13Mo: Final evaluation. Endocrine assessment. 24h Ambulatory BP measurement, anthropometric and metabolic evaluation. Quality of life and cognition questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 80 years.
* Unilateral SCSI:

  * Incidentally discovered adrenal tumor with attenuation < 20 UH and/or relative wash-out (> 40%) or absolute wash-out (> 60%) of contrast media and size ≥ 2 cm. Tumors that do not fulfil these criteria might be included if their size is ≤ 4 cm, do not exhibit signs of malignancy (necrosis areas, large and irregular rims) and are stable in size after ≥ 6 months of follow-up.
  * Impaired 1 mg dexamethasone suppression (Cortisol > 138 nmol/L or 5 µg/dL), OR Impaired 1 mg dexamethasone suppression (Cortisol > 50 nmol/L or 1.8 µg/dL) AND one biochemical abnormalities among:

    * 08h00 plasma ACTH < 2.2 pmol/L or plasma ACTH following CRH injection ≤ 6.6 pmol/L,
    * midnight plasma cortisol > 150 nmol/L,
    * increased late evening salivary cortisol,
    * UFC between 1 and 2.0 x N.
  * Treated BP (and confirmed using an automated home BP monitoring) OR increased BP (≥ 135/85 mmHg) none treated, using an automated home BP monitoring.

Exclusion Criteria:

* Age > 80 y,
* Bilateral SCSI, Warning: Contralateral nodular formations < 10 mm are considered as negligible,
* Incidentally discovered adrenal tumor size < 2 cm,
* Malignant hypertension, stroke, pulmonary oedema or myocardial infarction during the previous year,
* Malignant hypertension during the Run-in period,
* Obligatory beta blocker treatment. Patients receiving betablocker treatment for other purpose than hypertension can be included. However, to be included, patients should need at least an extrastep of hypertensive treatment in order to allow the SAHR decrease following randomisation. The dose of betablocker has to stay the same during all the study.
* UFC > ULN x 2.0 N,
* 8h00 plasma ACTH > 20 pg/ml (4.4 pmol/L),
* Chronic renal insufficiency (clearance < 30 mL/min)
* Dissipation of the biological endocrine criteria for SCSI at the end of the Run-In period,
* Intake of exogenous corticoids or drugs that interfere with dexamethasone metabolism,
* Pregnancy,
* Childbearing woman with no contraceptive effective method (HAS criteria - 77),
* Adverse pathological conditions responsible for reduced life expectancy.

Exclusion criteria after the Run-In period:

* Spontaneous resolution of biological features of SCSI
* Hypertension not confirmed with standard blood pressure self-measurement device
* Hypertension not controlled (≥ 135/85 mmHg) at the end of the Run-In period
* Malignant hypertension (> 175/115 mmHg)
* Patient receiving betablocker and not receiving at least an extrastep of hypertensive treatment of the SAHR

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Blood pressure value and SAHR step 12 months after inclusion | 13 months
  Treatment response will defined as a reduction of at least 1 step of SAHR at the end of the study, with BP maintained within the study objectives (<135 mm Hg systolic and <85 mm Hg diastolic) according to self-measurement at home.

SECONDARY OUTCOMES:
Antihypertensive treatment score and daily drug dose | 12 months
Incidence of complications in the two strategies. | 12 months
Direct costs of the two strategies. | 12 months
Assessment of predictive factors for the success of surgery on BP | 12 months
  age, family history of hypertension, duration of hypertension, kidney function, biochemical endocrine abnormalities, urinary steroid profile
number of patients requiring antihypertensive treatment | 12 months
24 hours ambulatory blood pressure monitoring values | At inclusion (day 0) and at 12 months
Blood glucose and lipid lowering agents values | 12 months
Cardiovascular risk factors/markers level | 12 months
  Comparison of the two therapeutic strategies with regard to cardiovascular risk factors/markers: BMI, body composition evaluated by DEXA, abdominal fat evaluated on CT-scan, fasting blood glucose and insulin, HbA1C, HOMA-IR (homeostasis model of assessment of insulin resistance) and OGTT (oral glucose tolerance test), blood lipids, pro-inflammatory adipokines
Number of patients with persistent diabetes, dyslipidemia and metabolic syndrome | 12 months
Evaluation of quality of life | At inclusion and 12 months
  Comparison of the two therapeutic strategies with regard to quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Eric FRISON, Dr, Study Chair — University Hospital, Bordeaux
Locations (17):
- France (14):
  - Service de Médecine Interne, Endocrinologie et Nutrition - CHU de Strasbourg, Strasbourg, Alsace
  - Service Endocrinologie, Diabétologie, maladies métaboliques - CHU de Bordeaux, Pessac, Aquitaine
  - Service d'Endocrinologie - Niveau 18 - Caen CHU Côte de Nacre, Caen, Basse-Normandie
  - Service d'Endocrinologie, Diabétologie, Nutrition - CHU d'Amiens, Amiens, Haut de France
  - Endocrinologie, Diabète et Maladies Métaboliques - CHU de Rouen, Rouen, Haute-Normandie
  - Service d'Endocrinologie, Diabétologie et Métabolisme - CHRU de LILLE, Lille, Hauts-de-France
  - Service d'Endocrinologie et Maladies Métabolique - CHU de Toulouse, Toulouse, Midi-Pyrénées
  - Département Endocrinologie-Diabétologie -Nutrition - CHU d'ANGERS, Angers, Pays de la Loire Region
  - CIC Endocrinologie-Nutrition - CHU de Nantes, Nantes, Pays de la Loire Region
  - Service d'Endocrinologie, Diabète et Maladies Métaboliques - Assistance publique - Hôpitaux de Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU de Poitiers, Poitiers
  - Service d'Endocrinologie et des Maladies de la Reproduction- Assistance Publique - Hôpitaux de Paris - Hôpial Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - Assistance Publique - Hôpitaux de Paris - Hôpital COCHIN, Paris, Île-de-France Region
  - Service d'Hypertension et de Médecine Vasculaire - Assistance Publique - Hôpitaux de Paris - Hôpital européen Georges Pompidou, Paris, Île-de-France Region
- Germany (2):
  - Endokrinologie, Diabetes und Ernährungsmedizin, Campus Mitte, Medizinische Klinik - Charité - Universitätsmedizin Berlin, Berlin
  - Department of Internal Medicine I, Endocrine and Diabetes Uni -University Hospital Würzburg, Würzburg
- S Orsola-Malpighi Hospital, Bologna, Italy

REFERENCES:
- [Derived] Tabarin A, Espiard S, Deutschbein T, Amar L, Vezzossi D, Di Dalmazi G, Reznik Y, Young J, Desailloud R, Goichot B, Drui D, Assie G, Lefebvre H, Mai K, Castinetti F, Laboureau S, Terzolo M, Ferriere A, Georget A, Frison E, Vantyghem MC, Fassnacht M, Gosse P; CHIRACIC Collaborators. Surgery for the treatment of arterial hypertension in patients with unilateral adrenal incidentalomas and mild autonomous cortisol secretion (CHIRACIC): a multicentre, open-label, superiority randomised controlled trial. Lancet Diabetes Endocrinol. 2025 Jul;13(7):580-590. doi: 10.1016/S2213-8587(25)00062-2. Epub 2025 May 12. PMID 40373786